CLINICAL TRIAL: NCT05205161
Title: A Modular Phase I/II, Open-label, Dose Escalation and Expansion, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of AZD0466 as Monotherapy or in Combination With Anticancer Agents in Patients With Advanced Non-Hodgkin Lymphoma.
Brief Title: A Phase I/II Study of AZD0466 as Monotherapy or in Combination With Anticancer Agents in Advanced Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to safety reasons.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8242C00001; 2021-003410-39 (EudraCT Number)
Record Dates: First submitted 2022-01-05; First posted 2022-01-25 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Open-label,; Dose Escalation; Dose Expansion,; Multicentre Study; Anticancer; Pegylated poly-L-lysine dendrimer
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — AZD0466

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part A (Dose Escalation): Dose Level (DL)-1 (Experimental): Participants with advanced R/R B-NHL will receive AZD0466 on day 1 , day 4, day 8 day 15, day 22 of cycle 1 and day 1, day 8 day 15, day 22 of cycle 2 and beyond until maximum 2 years or until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study intervention, whichever occurs first.
  Interventions: Drug: AZD0466
- Part A (Dose Escalation): DL1 (Experimental): Participants with advanced R/R B-NHL will receive AZD0466 on day 1 , day 4, day 8 day 15, day 22 of cycle 1 and day 1, day 8 day 15, day 22 of cycle 2 and beyond until maximum 2 years or until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study intervention, whichever occurs first.
  Interventions: Drug: AZD0466
- Part A (Dose Escalation): DL2 (Experimental): Participants with advanced R/R B-NHL will receive AZD0466 on day 1 , day 4, day 8 day 15, day 22 of cycle 1 and day 1, day 8 day 15, day 22 of cycle 2 and beyond until maximum 2 years or until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study intervention, whichever occurs first.
  Interventions: Drug: AZD0466
- Part A (Dose Escalation): DL3 (Experimental): Participants with advanced R/R B-NHL will receive AZD0466 on day 1 , day 4, day 8 day 15, day 22 of cycle 1 and day 1, day 8 day 15, day 22 of cycle 2 and beyond until maximum 2 years or until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study intervention, whichever occurs first.
  Interventions: Drug: AZD0466
- Part A (Dose Escalation): DL4 (Experimental): Participants with advanced R/R B-NHL will receive AZD0466 on day 1 , day 4, day 8 day 15, day 22 of cycle 1 and day 1, day 8 day 15, day 22 of cycle 2 and beyond until maximum 2 years or until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study intervention, whichever occurs first.
  Interventions: Drug: AZD0466
- Part B (Dose Expansion): Cohort B1 (R/R MCL) (Experimental): Participants with advanced R/R MCL will receive AZD0466 at the recommended phase 2 dose (RP2D) until maximum 2 years or until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study intervention, whichever occurs first.
  Interventions: Drug: AZD0466
- Part B (Dose Expansion): Cohort B2 (R/R FL or MZL) (Experimental): Participants with advanced R/R FL or MZL will receive AZD0466 at the recommended phase 2 dose (RP2D) until maximum 2 years or until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study intervention, whichever occurs first.
  Interventions: Drug: AZD0466
- Part B (Dose Expansion): Cohort B3 (R/R DLBCL) (Experimental): Participants with advanced R/R DLBCL will receive AZD0466 at the recommended phase 2 dose (RP2D) until maximum 2 years or until disease progression, initiation of alternative anticancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue study intervention, whichever occurs first.
  Interventions: Drug: AZD0466

INTERVENTIONS:
Drug: AZD0466 — All patients will receive treatment with the investigational product AZD0466 via intravenous infusion.

SUMMARY:
This study evaluates the safety, tolerability, PK, and preliminary efficacy of AZD0466 as monotherapy or in combination with other anticancer agents in patients with advanced NHL

DETAILED DESCRIPTION:
This is a modular Phase I/II, open-label, dose escalation and expansion, multicentre Study. The study consists of individual modules, each evaluating the safety and tolerability of AZD0466 as monotherapy or with a specific combination treatment. The initial components are the core protocol, which contains information applicable to all modules, and Module 1.

Module 1 will evaluate the safety, tolerability, PK, and preliminary efficacy of AZD0466 monotherapy and will include 2 parts. Part A dose escalation and Part B dose expansion cohorts. Part A will enrol patients with advanced B-NHL and once the RP2D has been determined, Part B may open to further explore the preliminary anticancer efficacy of AZD0466 monotherapy in patients with selected lymphoid malignancies.

Part A: Phase 1 dose setting to assess the safety and tolerability and determine dose(s) and schedule(s) to be evaluated in Part B.

Part B: Phase 1b/2a dose expansion to assess the efficacy of AZD0466 in 3 select patient populations: relapsed/refractory (R/R) mantle cell lymphoma (MCL) (Cohort B1), R/R follicular lymphoma (FL) or marginal zone lymphoma (MZL) (Cohort B2), and R/R diffuse large B-cell lymphoma (DLBCL) (Cohort B3).

ELIGIBILITY:
Inclusion Criteria- Core

* Patient must be aged ≥ 18 years at the time of signing the informed consent. In some countries, parental consent may be required in addition to an assent form for patients who are 18 years of age.
* Patient must have histologically documented diagnosis of B-cell non-Hodgkin lymphoma (B-NHL) as defined by a B-cell neoplasm in the World Health Organisation classification scheme except as noted in the exclusion criteria.
* Patient has relapsed after or failed to respond to at least 2 but no more than 5 prior systemic treatment regimens (including investigational therapy) and for whom there is no available therapy expected to improve survival (eg, standard chemotherapy, autologous stem cell transplantation (SCT), chimeric antigen receptor T cell (CAR-T) cell therapy).
* Documented active disease requiring treatment that is relapsed or refractory defined as:

  * Recurrence/relapse of disease after response to prior line(s) of therapy.
  * Progressive disease (refractory) on/after completion of the treatment regimen preceding entry into the study.
* Must have at least one measurable, fluorodeoxyglucose positron emission tomography (FDG-PET) avid lesion (except for MZL), based on bi-dimensional assessment on PET and computed tomography (CT)/magnetic resonance imaging (MRI) scan. A measurable lesion is defined as:

  * For nodal lesions: longest diameter > 1.5 cm
  * For extranodal lesions: longest diameter > 1 cm
* Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2. Performance status must not have deteriorated by ≥ 2 levels within 2 weeks after providing informed consent.
* Adequate haematologic, hepatic, and renal function
* Adequate cardiac function as demonstrated by left ventricular ejection fraction > 50% on screening cardiac multigated acquisition, magnetic resonance imaging, or echocardiogram.
* Women of childbearing potential and men should use protocol defined contraceptive measures.
* Willing and able to participate in all required study evaluations and procedures including receiving IV administration of study intervention and admission to the hospital, when required, for administration of study treatment and monitoring.
* All patients must be willing to undergo an incisional or excisional lymph node or tissue biopsy or to provide a lymph node or tissue biopsy from the most recent available archival tissue.
* For inclusion in the genetic component of the study, patients must fulfil protocol defined criteria.

Inclusion Criteria- Module 1

Additional Inclusion Criteria for Cohort B1 (R/R mantle cell lymphoma [MCL]):

* Histologically confirmed MCL, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1, as assessed by Investigator or local pathologist.
* Must have relapsed after or failed to respond to at least 2 prior lines of treatment, including one anti-CD20 monoclonal antibody (mAb) and a Bruton's tyrosine kinase inhibitor.

Additional Inclusion Criteria for Cohort B2 (R/R FL or MZL):

* Histologically confirmed diagnosis of FL Grade 1, 2, or 3a OR histologically confirmed MZL including splenic, nodal, and extranodal subtypes, as assessed by Investigator or local pathologist.
* For FL patients: Previously received at least 2 prior systemic treatment regimens (including anti-CD20 mAb and an alkylating agent).
* For MZL patients: Previously received at least 2 prior lines of systemic therapy including at least one anti-CD20 mAb-directed regimen either as monotherapy or as chemoimmunotherapy (Helicobacter pylori eradication and radiation therapy alone will not be considered a systemic treatment regimen).

Additional Inclusion Criteria for Cohort B3 (R/R DLBCL):

* Histologically confirmed DLBCL (including transformed FL) OR FL Grade 3b.
* Must have received 2 lines of systemic therapy including at least one anti-CD20 mAb-directed regimen and must have failed or are ineligible for stem cell transplantation (if indicated per local institutional guidelines).

Exclusion Criteria- Core

* Diagnosis of post-transplant lymphoproliferative disease, Richter's transformation, Burkitt's lymphoma, Burkitt-like lymphoma, lymphoblastic lymphoma/leukaemia, chronic lymphocytic leukaemia, small lymphocytic lymphoma.
* High risk of TLS according to Howard modification of Cairo-Bishop criteria and/or the presence of bulky disease.
* Unresolved toxicity from prior anticancer therapy. Patients with Grade 2 neuropathy or Grade 2 alopecia are eligible.
* Active idiopathic thrombocytopenic purpura.
* Active central nervous system (CNS) involvement by lymphoma, leptomeningeal disease or spinal cord compression.
* Known history of infection with human immunodeficiency virus.
* Known serologic status reflecting active hepatitis B or C infection; concurrent infection with cytomegalovirus (CMV).
* Patients must be tested for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and those with active infection in accordance with local testing guidelines will be excluded.
* Any evidence of severe or uncontrolled systemic diseases; current unstable or uncompensated respiratory or cardiac conditions; uncontrolled hypertension; history of, or active, bleeding diatheses; uncontrolled active systemic fungal, bacterial, or other infection.
* Any of the following cardiac criteria at screening: patients with a history of myocarditis within one year of study entry, or heart failure; mean resting corrected QT interval (QTcF) ≥ 470 msec obtained from 3 electrocardiograms (ECGs), in the absence of a cardiac pacemaker; any factors that increase the risk of QTc prolongation or risk of arrhythmic events; any clinically important abnormalities in rhythm, conduction or morphology of resting ECG.
* History of another life-threatening malignancy ≤ 2 years prior to first dose of study intervention.
* Any of the following currently or in the 6 months prior to the first dose of study intervention: coronary artery bypass graft; angioplasty; vascular stent; myocardial infarction; angina pectoris; haemorrhagic or thrombotic stroke, including transient ischaemic attacks or any other CNS bleeding.
* Treatment with any of the following: radiotherapy less than 2 weeks prior to the first dose of study intervention; any investigational agents or study drugs from a previous clinical study within ≤ 14 days or 5 half-lives prior to the first dose of study intervention; any other chemotherapy, immunotherapy, immunosuppressant medication or anticancer agents within 21 days of the first dose of study intervention; Prior allogenic haematopoietic stem cell transplantation (HSCT) within 6 months from the first dose of study intervention (patients > 6 months after allogenic HSCT are eligible in the absence of active graft-versus host disease and concomitant immune-suppressive therapy). Eligible patients must have stopped immunosuppression at least 2 months prior to study entry; prior cellular therapies such as CAR-T and/or autologous HSCT within 3 months prior to the first dose of study intervention; major surgery ≤ 21 days, or minor surgical procedures ≤ 7 days, prior to the first dose of study intervention; prescription or non-prescription drugs or other products known to be sensitive substrates of BCRP, OCT2, OAT3, OATP1B1, OATP1B3, CYP2B6, CYP2C8, CYP2C9 or CYP2D6, or reversible moderate or strong cytochrome 3A (CYP3A) inhibitors, which cannot be discontinued within 5 half-lives of the first dose of study intervention and withheld throughout the study until 14 days after the last dose of AZD0466; moderate or strong mechanism-based inhibitors or inducers of CYP3A4 which cannot be discontinued within 5 half-lives plus 12 days of the drug prior to the first dose of study intervention and withheld until 14 days after the last dose of AZD0466; concurrent anticoagulation therapy, including aspirin, which cannot be stopped; medications with known risk of Torsades de Pointes within 5 half-lives of the first dose of study intervention and continuing until 5 half-lives after the last dose of AZD0466.
* Administration of a live, attenuated vaccine within 4 weeks before first dose of study intervention.
* Administration of inactivated vaccines or protein/RNA immunogen vaccines.
* Patients with a known hypersensitivity to polyethylene glycol, pegylated products, or drugs with a similar chemical structure or class to AZD0466 or other BH3 mimetic.

Exclusion Criteria- Module 1

Additional Exclusion Criteria for Cohort B1:

- Patients with known blastoid or pleiomorphic variant at study entry/most recent relapse.

Additional Exclusion Criteria for Cohort B2:

* Histologically confirmed diagnosis of FL grade 3B.
* Known transformation to aggressive lymphoma, eg, large cell lymphoma.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Research Site, Duarte, California, United States
- Research Site, Heidelberg, Australia
- Research Site, Lille, France
- Research Site, Milan, Italy
- Research Site, Porto, Portugal
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D8242C00001_CSP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8242C00001&attachmentIdentifier=01178919-abc6-4791-bd50-907b6aa818c2&fileName=D8242C00001_CSP_Redacted.pdf&versionIdentifier=
- See also: D8242C00001_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8242C00001&attachmentIdentifier=976eceb2-efb8-4299-b4e0-177f19b7f1ff&fileName=D8242C00001_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: D8242C00001_SAP_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8242C00001&attachmentIdentifier=71a56b23-b13c-47ce-b026-ba1b035ed192&fileName=D8242C00001_SAP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study from 05July 2022 (First subject in) to 17 August 2023 (Last subject last visit) at 24 sites in 8 countries.
Pre-assignment Details: Participants meeting the inclusion criteria were enrolled in the study. All the assessments were performed as per the schedule of the assessments.
Groups:
- 600 mg of AZD0466: Participants received 600mg of AZ0466 in Part A of the treatment
- 1200 mg of AZD0466: Participants received 1200 mg of AZD0466 in Part A of the treatment
- 2400 mg of AZD0466: Participants received 2400mg of AZD0466 in Part A of the treatment
Period: Overall Study
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Started | 3 | 3 | 1
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 1
Not completed — Study terminated by sponsor | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- 1200 mg of AZD0466: Participants received 1200mg of AZD0466 in Part A of the treatment
- Total: Total of all reporting groups
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466 | Total
Number analyzed (Participants) | 3 | 3 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (7.0) | 44.0 (16.1) | NA (NA) — Since there is 1 participant, therefore descriptive statistics like mean and SD cannot be calculated | 57.0 (16.9)
Sex/Gender, Customized [Number; unit: Participants] — For Single participant in a particular gender, the data was not reported under specific gender, rather customised option was used, and the data was reported as Other to maintain participant's confidentiality
  Participants
    Male | 3 | 2 | 0 | 5
    Female | 0 | 0 | 0 | 0
    Other | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: Participants] — For Single participant in a particular race, the data was not reported under specific race, rather customised option was used, and the data was reported as Other to maintain participant's confidentiality
  Participants
    Asian | 2 | 0 | 0 | 2
    White | 0 | 2 | 0 | 2
    Not Reported | 0 | 1 | 0 | 1
    Other | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Number; unit: Participants] — For Single participant in a particular ethnic group, the data was not reported under specific ethnicity, rather customised option was used, and the data was reported as Other to maintain participant's confidentiality
  Participants
    Not Hispanic or Latino | 3 | 2 | 0 | 5
    Not Reported | 0 | 1 | 0 | 1
    Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE)
Description: The safety and the tolerability of AZD0466 in patients with relapsed/ refractory B-cell non-Hodgkin lymphoma (R/R B-NHL) was evaluated.
Time Frame: Day 1 to Follow-up (30 days post last dose or up to the day prior to start of subsequent cancer therapy) up to approximately 1 year 1 month
Population: The safety analysis included all participants who received at least one dose of AZD0466.
Measure: Number; unit: Participants
Groups:
- 600mg of AZD0466: Participants received 600 mg of AZ0466 in Part A of the treatment
- 2400 mg of AZD0466: Participants received 2400 mg of AZD0466 in Part A of the treatment
Arm/Group | 600mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
Participants
  Any AE | 3 | 3 | 1
  Any possibly related AE | 2 | 3 | 1
  Any AE of >= CTCAE grade 3 | 1 | 2 | 1
  Any Serious Adverse events (SAE) | 0 | 0 | 1
  Any possibly related SAE | 0 | 0 | 1
  Any SAE with outcome death | 0 | 0 | 0
  Any SAE of >= CTCAE grade 3 | 0 | 0 | 1
  Any Adverse event of Special interest | 0 | 1 | 0
  Any AE leading to discontinuation of AZD0466 | 0 | 1 | 1
  Any AE leading to AZD0466 drug interruption | 0 | 0 | 0
  Any AE leading to AZD0466 dose reduction | 0 | 0 | 0
  Any possibly related deaths | 0 | 0 | 0

2. Secondary Outcome: Part A: Maximum Observed Plasma (Peak) Drug Concentration (Cmax) of AZD4320
Description: The Cmax of AZD4320 was assessed to characterise the pharmacokinetic (PK) profile of AZD0466.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1
Population: The Pk analysis set included dosed participants with reportable plasma concentrations and no important AEs or protocol deviations that may impact Pk.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
nmol/L
  Total AZD4320 (Cycle 1 Day 8) | 46860 (11820) | 77090 (28580) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the Statistical Analysis Plan (SAP).
  Total AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Total AZD4320 (Cycle 2 Day 1) | 47970 (13460) | 72620 (26820) |
  Released AZD4320 (Cycle 1 Day 8) | 1035 (619.4) | 3658 (5033) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Released AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Released AZD4320 (Cycle 2 Day 1) | 585.9 (345.7) | 1760 (2174) |

3. Secondary Outcome: Part A: Time to Reach Peak or Maximum Observed Concentration or Response Following Drug Administration (Tmax) of AZD4320
Description: The tmax of AZD4320 was assessed to characterise the Pk profile of AZD0466.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Groups:
- 600 mg of AZD0466: Participants received 600 mg of AZ0466 in Part A of the treatment
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
hour
  Total AZD4320 (Cycle 1 Day 8) | 1.133 [0.67 to 1.23] | 1.083 [1.00 to 1.52] | NA [NA to NA] — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Total AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Total AZD4320 (Cycle 2 Day 1) | 1.917 [1.12 to 2.08] | 1.167 [1.00 to 2.03] |
  Released AZD4320 (Cycle 1 Day 8) | 1.167 [1.13 to 1.23] | 2.017 [2.00 to 2.12] | NA [NA to NA] — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Released AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Released AZD4320 (Cycle 2 Day 1) | 1.12 [1.12 to 1.17] | 2.033 [2.00 to 2.10] |

4. Secondary Outcome: Part A: Terminal Rate Constant, Estimated by Log-linear Least Squares Regression of the Terminal Part of the Concentration-time Curve (λz) of AZD4320
Description: The λz of AZD4320 was assessed to characterise the Pk profile of AZD0466.
Time Frame: Cycle 1 Day 8 (Study Day 8), Cycle 2 Day 1 (Study Day 22)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
1/hour
  Total AZD4320 (Cycle 1 Day 8) | 0.05729 (0.003854) | 0.06054 (0.005678) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Total AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Total AZD4320 (Cycle 2 Day 1) | 0.06238 (0.01430) | 0.06157 (0.008283) |
  Released AZD4320 (Cycle 1 Day 8) | 0.02643 (0.006131) | 0.03251 (0.008458) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Released AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 2 | 2 | 0
  Released AZD4320 (Cycle 2 Day 1) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP. | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP. |

5. Secondary Outcome: Part A: Half-life Associated With Terminal Slope (λz) of a Semi-logarithmic Concentration-time Curve (t1/2λz) of AZD4320
Description: The t1/2λz of AZD4320 was assessed to characterise Pk profile of AZD0466.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
hour
  Total AZD4320 (Cycle 1 Day 8) | 12.14 (0.8454) | 11.52 (1.062) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Total AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Total AZD4320 (Cycle 2 Day 1) | 11.48 (2.389) | 11.39 (1.515) |
  Released AZD4320 (Cycle 1 Day 8) | 27.35 (7.302) | 22.22 (5.234) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Released AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 2 | 2 | 0
  Released AZD4320 (Cycle 2 Day 1) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP. | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP. |

6. Secondary Outcome: Part A: Partial Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours After the Start of Infusion (AUC0-24) of AZD4320
Description: The AUC0-24 of AZD4320 was assessed to characterise the Pk profile of AZD0466.
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
h*nmol/L
  Total AZD4320 (Cycle 1 Day 8) | 429900 (143900) | 736800 (405900) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Total AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Total AZD4320 (Cycle 2 Day 1) | 479200 (204200) | 660700 (388900) |
  Released AZD4320 (Cycle 1 Day 8) | 7112 (4377) | 30340 (40570) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Released AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 2 | 2 | 0
  Released AZD4320 (Cycle 2 Day 1) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP. | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP. |

7. Secondary Outcome: Part A: Partial Area Under the Plasma Concentration-time Curve From Time 0 to 72 Hours After the Start of Infusion (AUC0-72) of AZD4320
Description: The AUC0-72 of AZD4320 was assessed to characterise the Pk profile of AZD0466.
Time Frame: Cycle 1 Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
h*nmol/L
  Total AZD4320 (Cycle 1 Day 8) | 565200 (193800) | 930500 (543900) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Released AZD4320 (Cycle 1 Day 8) | 13320 (8190) | 36710 (42900) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.

8. Secondary Outcome: Part A: Area Under the Plasma Concentration-curve From Time 0 to the Last Quantifiable Concentration (AUClast) of AZD4320
Description: The AUClast of AZD4320 was assessed to characterise the Pk profile of AZD0466
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
h*nmol/L
  Total AZD4320 (Cycle 1 Day 8) | 566000 (190300) | 930200 (543800) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Total AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Total AZD4320 (Cycle 2 Day 1) | 473600 (204500) | 634800 (360600) |
  Released AZD4320 (Cycle 1 Day 8) | 12800 (8628) | 36690 (42910) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Released AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Released AZD4320 (Cycle 2 Day 1) | 6616 (3688) | 18520 (22660) |

9. Secondary Outcome: Part A: Time of Last Observed (Quantifiable) Concentration (Tlast) of AZD4320
Description: The tlast of AZD4320 was assessed to characterise the Pk profile of AZD0466
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
hour
  Total AZD4320 (Cycle 1 Day 8) | 72.117 [69.05 to 95.87] | 71.683 [70.93 to 71.75] | NA [NA to NA] — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Total AZD430 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Total AZD430 (Cycle 2 Day 1) | 23.233 [22.10 to 24.22] | 22.333 [22.00 to 23.50] |
  Released AZD4320 (Cycle 1 Day 8) | 1.167 [1.13 to 1.23] | 2.017 [2.00 to 2.12] | NA [NA to NA] — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Released AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Released AZD4320 (Cycle 2 Day 1) | 23.233 [22.10 to 24.22] | 22.333 [22.00 to 23.50] |

10. Secondary Outcome: Part A: Concentration Prior to Dosing (Ctrough) of AZD4320
Description: The Ctrough of AZD4320 was assessed to characterise the Pk profile of AZD0466
Time Frame: Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 0
nmol/L
  Total AZD430 (Cycle 2 Day 1): number analyzed (Participants) | 2 | 3 | 0
  Total AZD430 (Cycle 2 Day 1) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP. | 48.80 (43.96) |
  Released AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 2 | 3 | 0
  Released AZD4320 (Cycle 2 Day 1) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP. | 2.277 (2.145) |

11. Secondary Outcome: Part A:Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Quantifiable Analyte Concentration Divided by the Dose Administered (Dose Normalised AUClast) of AZD4320
Description: The Dose normalised AUClast of total AZD4320 was assessed to characterise the Pk profile of AZD0466
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*nmol/L/mg
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
h*nmol/L/mg
  Total AZD430 (Cycle 1 Day 8) | 943.4 (317.2) | 775.1 (453.2) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Total AZD430 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Total AZD430 (Cycle 2 Day 1) | 789.4 (340.8) | 529.0 (300.5) |

12. Secondary Outcome: Part A: Area Under the Plasma Concentration-time Curve From Time 0 to 72 Hours After the Start of Infusion (Dose Normalised AUC0-72) of AZD4320
Description: The Dose normalised AUC0-72 of total AZD4320 was assessed to characterise the Pk profile of AZD0466
Time Frame: Cycle 1 Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*nmol/L/mg
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
h*nmol/L/mg | 942.0 (323.0) | 775.4 (453.3) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.

13. Secondary Outcome: Part A: Maximum Observed Plasma (Peak) Drug Concentration Divided by the Dose Administered (Dose Normalised Cmax) of AZD4320
Description: The Dose normalised Cmax of total AZD4320 was assessed to characterise the Pk profile of AZD0466
Time Frame: Cycle 1 Day 8, Cycle 2 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nmol/L/mg
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
nmol/L/mg
  Total AZD4320 (Cycle 1 Day 8) | 78.11 (19.70) | 64.24 (23.81) | NA (NA) — Due to insufficient number of participants (less than 3), no summary statistics were presented as per methodology mentioned in the SAP.
  Total AZD4320 (Cycle 2 Day 1): number analyzed (Participants) | 3 | 3 | 0
  Total AZD4320 (Cycle 2 Day 1) | 79.95 (22.44) | 60.51 (22.35) |

14. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: The DLT of AZD0466 in participants with R/R B-NHL was evaluated.
Time Frame: Day 1 to end of Cycle 1 (28 days treatment cycle)
Population: The safety analysis included all participants who received at least one dose of AZD0466.
Measure: Number; unit: Participants
Arm/Group | 600 mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
Number analyzed (Participants) | 3 | 3 | 1
Participants | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Follow-up (30 days post last dose or up to the day prior to start of subsequent cancer therapy) up to approximately 1 year 1 month
Arm/Group | 600mg of AZD0466 | 1200 mg of AZD0466 | 2400 mg of AZD0466
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 600mg of AZD0466 (N=3) | 1200 mg of AZD0466 (N=3) | 2400 mg of AZD0466 (N=1)
Troponin increased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 600mg of AZD0466 (N=3) | 1200 mg of AZD0466 (N=3) | 2400 mg of AZD0466 (N=1)
COVID-19 (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Discomfort (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0
Platelet count decreased (Investigations) | 2 | 2 | 0

LIMITATIONS AND CAVEATS:
In this study, no participants were enrolled/screened in Module 1 Part B of this study, thus only results from Module 1 Part A will be presented in the report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No unpublished information contained herein may be disclosed without prior written approval from AstraZeneca AB. Access to this document must be restricted to relevant parties.

DOCUMENTS (2):
  • Study Protocol (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT05205161/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT05205161/SAP_001.pdf